CLINICAL TRIAL: NCT00955877
Title: Randomized, Double-Blinded Placebo Controlled Trial of Epidural, Sustained-relief Morphine for Acute Post-operative Analgesia Following Selective Dorsal Rhizotomy in Children
Brief Title: Extended-release Epidural Morphine for Acute Post-operative Analgesia Following Selective Dorsal Rhizotomy in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The manufacturer decided to stop drug production.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DeporDur2009
Record Dates: First submitted 2009-08-03; First posted 2009-08-10 (Estimated); Results first posted 2018-06-13 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Spastic Cerebral Palsy
Keywords: extended-release epidural morphine; DepoDur; Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DepoDur80 (Experimental): DepoDur will be administered at 80μg/kg (not to exceed 5 mg total/patient) under direct vision in the L1 laminectomy defect prior to wound closure.
  Interventions: Drug: Extended-release Epidural morphine (EREM) 80
- DepoDur120 (Experimental): DepoDur will be administered at 120μg/kg (not to exceed 10 mg total/patient) under direct vision in the L1 laminectomy defect prior to wound closure.
  Interventions: Drug: Extended-release Epidural Morphine (EREM) 120
- Control (Placebo Comparator): Preservative-free normal saline (2.5ml) will be placed in the L1 laminectomy defect and also dispensed 1-2 levels above and 1-2 levels below using a flexible angiocatheter prior to wound closure.
  Interventions: Drug: Control: Saline

INTERVENTIONS:
Drug: Extended-release Epidural morphine (EREM) 80 — After completion of the rhizotomy, the dura will be closed in the standard water-tight fashion with running suture. Epidural DepoDur (80μg/kg) will be placed under direct vision in the L1 laminectomy defect. It will also be dispensed 1-2 levels above and 1-2 levels below using a flexible angiocatheter.
  Other Names: DepoDur
  Arms: DepoDur80
Drug: Extended-release Epidural Morphine (EREM) 120 — After completion of the rhizotomy, the dura will be closed in the standard water-tight fashion with running suture. Epidural DepoDur (120μg/kg) will be placed under direct vision in the L1 laminectomy defect. It will also be dispensed 1-2 levels above and 1-2 levels below using a flexible angiocatheter.
  Other Names: DepoDur
  Arms: DepoDur120
Drug: Control: Saline — After completion of the rhizotomy, the dura will be closed in the standard water-tight fashion with running suture. Preservative-free normal saline (2.5 ml) will be placed under direct vision in the L1 laminectomy defect. It will also be dispensed 1-2 levels above and 1-2 levels below using a flexible angiocatheter.
  Arms: Control

SUMMARY:
The purpose of this proposal is to improve the investigators' current Selective Dorsal Rhizotomy (SDR) analgesia protocol by eliminating or minimizing the use of fentanyl in the post-operative period.

Children undergoing SDR for spastic cerebral palsy have significant post-operative pain. The procedure requires dissection of the lumbar back musculature and removal of the L1 lamina (the bony posterior part of the vertebra). The majority of the operation is intradural, and a water-tight dural closure at the termination of the operation is critical in order to prevent leakage of cerebrospinal fluid (CSF) from the wound. In fact, these children must remain flat on their back for 48 hours to allow the dural incision to heal prior to mobilization. Thus, adequate pain control is essential not only for patient comfort, but also to prevent agitation and additional stress on the dural closure.

Currently, the investigators' patients undergoing SDR are treated for 48 hours with scheduled intravenous (IV) narcotic (continuous fentanyl infusion at 0.5-2.0 μg/kg/hour) in addition to the sedative/muscle relaxant Valium (0.2 mg/kg IV every 4 hours for 24 hours, then every 6 hours for 24 hours). The IV fentanyl, and to a lesser degree Valium, carries a real risk of hypotension and respiratory depression and requires frequent dose adjustments to achieve adequate analgesia.

By improving the current SDR analgesia protocol, the investigators hope to maximize patient safety and comfort while maintaining the effectiveness of the operation by minimizing the risk of CSF leak.

DETAILED DESCRIPTION:
improve the investigators' current Selective Dorsal Rhizotomy (SDR) analgesia protocol by eliminating or minimizing the use of fentanyl in the post-operative period.

Children undergoing SDR for spastic cerebral palsy have significant post-operative pain. The procedure requires dissection of the lumbar back musculature and removal of the L1 lamina (the bony posterior part of the vertebra). The majority of the operation is intradural, and a water-tight dural closure at the termination of the operation is critical in order to prevent leakage of cerebrospinal fluid (CSF) from the wound. In fact, these children must remain flat on their back for 48 hours to allow the dural incision to heal prior to mobilization. Thus, adequate pain control is essential not only for patient comfort, but also to prevent agitation and additional stress on the dural closure.

Currently, the investigators' patients undergoing SDR are treated for 48 hours with scheduled intravenous (IV) narcotic (continuous fentanyl infusion at 0.5-2.0 μg/kg/hour) in addition to the sedative/muscle relaxant Valium (0.2 mg/kg IV every 4 hours for 24 hours, then every 6 hours for 24 hours). The IV fentanyl, and to a lesser degree Valium, carries a real risk of hypotension and respiratory depression and requires frequent dose adjustments to achieve adequate analgesia.

By improving the current SDR analgesia protocol, the investigators hope to maximize patient safety and comfort while maintaining the effectiveness of the operation by minimizing the risk of CSF leak.

ELIGIBILITY:
Inclusion Criteria:

* Receiving selective dorsal rhizotomy (SDR)
* Willingness to Participate

Exclusion Criteria:

* Known Morphine Allergy
* Inability to speak and read the English language

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2010-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Limbrick, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Clark SL, Hankins GD. Temporal and demographic trends in cerebral palsy--fact and fiction. Am J Obstet Gynecol. 2003 Mar;188(3):628-33. doi: 10.1067/mob.2003.204. PMID 12634632
- [Background] Kuban KC, Leviton A. Cerebral palsy. N Engl J Med. 1994 Jan 20;330(3):188-95. doi: 10.1056/NEJM199401203300308. No abstract available. PMID 8264743
- [Background] Grether JK, Cummins SK, Nelson KB. The California Cerebral Palsy Project. Paediatr Perinat Epidemiol. 1992 Jul;6(3):339-51. doi: 10.1111/j.1365-3016.1992.tb00774.x. PMID 1635884
- [Background] Taft LT. Cerebral palsy. Pediatr Rev. 1995 Nov;16(11):411-8; quiz 418. No abstract available. PMID 8539191
- [Background] Steinbok P. Outcomes after selective dorsal rhizotomy for spastic cerebral palsy. Childs Nerv Syst. 2001 Jan;17(1-2):1-18. doi: 10.1007/pl00013722. PMID 11219613
- [Background] McLaughlin J, Bjornson K, Temkin N, Steinbok P, Wright V, Reiner A, Roberts T, Drake J, O'Donnell M, Rosenbaum P, Barber J, Ferrel A. Selective dorsal rhizotomy: meta-analysis of three randomized controlled trials. Dev Med Child Neurol. 2002 Jan;44(1):17-25. doi: 10.1017/s0012162201001608. PMID 11811645
- [Background] Wright FV, Sheil EM, Drake JM, Wedge JH, Naumann S. Evaluation of selective dorsal rhizotomy for the reduction of spasticity in cerebral palsy: a randomized controlled tria. Dev Med Child Neurol. 1998 Apr;40(4):239-47. doi: 10.1111/j.1469-8749.1998.tb15456.x. PMID 9593495
- [Background] Steinbok P, Reiner AM, Beauchamp R, Armstrong RW, Cochrane DD, Kestle J. A randomized clinical trial to compare selective posterior rhizotomy plus physiotherapy with physiotherapy alone in children with spastic diplegic cerebral palsy. Dev Med Child Neurol. 1997 Mar;39(3):178-84. doi: 10.1111/j.1469-8749.1997.tb07407.x. PMID 9112967
- [Background] McLaughlin JF, Bjornson KF, Astley SJ, Graubert C, Hays RM, Roberts TS, Price R, Temkin N. Selective dorsal rhizotomy: efficacy and safety in an investigator-masked randomized clinical trial. Dev Med Child Neurol. 1998 Apr;40(4):220-32. doi: 10.1111/j.1469-8749.1998.tb15454.x. PMID 9593493
- [Background] Chicoine MR, Park TS, Kaufman BA. Selective dorsal rhizotomy and rates of orthopedic surgery in children with spastic cerebral palsy. J Neurosurg. 1997 Jan;86(1):34-9. doi: 10.3171/jns.1997.86.1.0034. PMID 8988079
- [Background] Park TS, Johnston JM. Surgical techniques of selective dorsal rhizotomy for spastic cerebral palsy. Technical note. Neurosurg Focus. 2006 Aug 15;21(2):e7. PMID 16918228
- [Background] Hartrick CT, Hartrick KA. Extended-release epidural morphine (DepoDur): review and safety analysis. Expert Rev Neurother. 2008 Nov;8(11):1641-8. doi: 10.1586/14737175.8.11.1641. PMID 18986234
- [Background] Gambling D, Hughes T, Martin G, Horton W, Manvelian G; Single-Dose EREM Study Group. A comparison of Depodur, a novel, single-dose extended-release epidural morphine, with standard epidural morphine for pain relief after lower abdominal surgery. Anesth Analg. 2005 Apr;100(4):1065-1074. doi: 10.1213/01.ANE.0000145009.03574.78. PMID 15781524
- [Background] Carvalho B, Riley E, Cohen SE, Gambling D, Palmer C, Huffnagle HJ, Polley L, Muir H, Segal S, Lihou C, Manvelian G; DepoDur Study Group. Single-dose, sustained-release epidural morphine in the management of postoperative pain after elective cesarean delivery: results of a multicenter randomized controlled study. Anesth Analg. 2005 Apr;100(4):1150-1158. doi: 10.1213/01.ANE.0000149544.58230.FF. PMID 15781537
- [Background] Carvalho B, Roland LM, Chu LF, Campitelli VA 3rd, Riley ET. Single-dose, extended-release epidural morphine (DepoDur) compared to conventional epidural morphine for post-cesarean pain. Anesth Analg. 2007 Jul;105(1):176-83. doi: 10.1213/01.ane.0000265533.13477.26. PMID 17578973
- [Background] Viscusi ER, Martin G, Hartrick CT, Singla N, Manvelian G; EREM Study Group. Forty-eight hours of postoperative pain relief after total hip arthroplasty with a novel, extended-release epidural morphine formulation. Anesthesiology. 2005 May;102(5):1014-22. doi: 10.1097/00000542-200505000-00022. PMID 15851890
- [Background] Hartrick CT, Martin G, Kantor G, Koncelik J, Manvelian G. Evaluation of a single-dose, extended-release epidural morphine formulation for pain after knee arthroplasty. J Bone Joint Surg Am. 2006 Feb;88(2):273-81. doi: 10.2106/JBJS.D.02738. PMID 16452737
- [Background] Martin G, Hartmannsgruber M, Riley E, Manvelian G. Single-dose extended-release epidural morphine for pain after hip arthroplasty. J Opioid Manag. 2006 Jul-Aug;2(4):209-18. doi: 10.5055/jom.2006.0033. PMID 17319482
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163
- [Background] Jensen MP, Turner JA, Romano JM. Correlates of improvement in multidisciplinary treatment of chronic pain. J Consult Clin Psychol. 1994 Feb;62(1):172-9. doi: 10.1037//0022-006x.62.1.172. PMID 8034820
- [Background] Solodiuk J, Curley MA. Pain assessment in nonverbal children with severe cognitive impairments: the Individualized Numeric Rating Scale (INRS). J Pediatr Nurs. 2003 Aug;18(4):295-9. doi: 10.1016/s0882-5963(03)00090-3. PMID 12923744

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DepoDur80 | DepoDur120 | Control
Started | 6 (Drug manufacturer ceased producing the drug prior to completion of 10 enrolled in this arm.) | 0 (No patients were enrolled because analysis of previous arm wasn't completed.) | 7
Completed | 6 | 0 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DepoDur80 | DepoDur120 | Control | Total
Number analyzed (Participants) | 6 | 0 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 0 | 7 | 13
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 5 | 0 | 6 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 |  | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Adequacy of Analgesia as Judged by Age-adjusted Pain Scales
Description: Mean and standard deviation for standardized, age-appropriate pain scales (per patient per day) 48hrs post surgery. As is standard of care at St. Louis Children's Hospital, pain level was scored based on age using the "Face, Legs, Activity, Cry, Consolability" (FLACC) for participants aged 0-3, the FACES scale on participants between the age of 3 and 5, numeric pain rating scale (NRS) on participants between the age of 5 and 8 years, or the Individualized Numeric Rating Scale (INRS) for participants greater than or equal to 8 years of age. All four of the scales were ranged from 0-10 scores, with 0 being no pain at all, and 10 being extreme pain. Each patient had two scores given, one at 24hrs and one at 48hrs post surgery. The output was reported as an average of all scores for all patients within each group.
Time Frame: 48 hour post-operative period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DepoDur80 | DepoDur120 | Control
Number analyzed (Participants) | 6 | 0 | 7
units on a scale | 0.5454 (1.2136) |  | 1.8571 (1.8337)

2. Primary Outcome: Quantity of Fentanyl Administered
Description: Mean and standard deviation of total quantity of fentanyl administered (per patient per day) 48hrs post surgery.
Time Frame: 48 hour post-operative period
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | DepoDur80 | DepoDur120 | Control
Number analyzed (Participants) | 6 | 0 | 7
mcg | 11 (15.5037) |  | 10.7857 (10.6423)

3. Secondary Outcome: Number of Participants With Respiratory Depression Within 48hrs Post op
Description: Number of participants with respiratory depression within 48hrs post operation
Time Frame: 48 hour post-operative period
Measure: Count of Participants; unit: Participants
Arm/Group | DepoDur80 | DepoDur120 | Control
Number analyzed (Participants) | 6 | 0 | 7
Participants | 0 |  | 0

4. Secondary Outcome: Number of Participants With Hemodynamic Instability 48hrs Post op
Description: Number of Participants with Hemodynamic Instability 48hrs post operation
Time Frame: 48 hour post-operative period
Measure: Count of Participants; unit: Participants
Arm/Group | DepoDur80 | DepoDur120 | Control
Number analyzed (Participants) | 6 | 0 | 7
Participants | 0 |  | 0

5. Secondary Outcome: Number of Participants With CSF Leaks Within 6 Months Post op.
Description: Number of participants with CSF leaks within 6 months post operation.
Time Frame: 6 month post-operative period
Measure: Count of Participants; unit: Participants
Arm/Group | DepoDur80 | DepoDur120 | Control
Number analyzed (Participants) | 6 | 0 | 7
Participants | 0 |  | 0

6. Secondary Outcome: Number of Participants That Had Urine Retention for 48hrs Post Foley Catheter Removal.
Description: Number of participants that had urine retention for 48hrs post foley catheter removal.
Time Frame: After the Foley catheter has been removed on post-operative day #1 for a 48 hour follow-up period
Measure: Count of Participants; unit: Participants
Arm/Group | DepoDur80 | DepoDur120 | Control
Number analyzed (Participants) | 6 | 0 | 7
Participants | 0 |  | 0

7. Secondary Outcome: Number of Participants With Nausea and/or Vomiting 48hrs Post op.
Description: Number of participants with nausea and or vomiting 48hr post surgery
Time Frame: 48 hour post-operative period
Measure: Count of Participants; unit: Participants
Arm/Group | DepoDur80 | DepoDur120 | Control
Number analyzed (Participants) | 6 | 0 | 7
Participants | 6 | 0 | 6

8. Secondary Outcome: Number of Participants With Pruritis Within 48hrs Post op
Description: Number of participants with pruritis within 48hrs post operation
Time Frame: 48 hour post-operative period
Measure: Count of Participants; unit: Participants
Arm/Group | DepoDur80 | DepoDur120 | Control
Number analyzed (Participants) | 6 | 0 | 7
Participants | 2 |  | 0

9. Secondary Outcome: Number of Participants That Were Given Codeine 48hr Post Surgery
Description: Number of participants that were given codeine 48hr post surgery
Time Frame: 48hr post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | DepoDur80 | DepoDur120 | Control
Number analyzed (Participants) | 6 | 0 | 7
Participants | 1 |  | 2

10. Secondary Outcome: Number of Participants That Were Given Zofran 48hr Post Surgery
Description: Number of participants that were given Zofran 48hr post surgery
Time Frame: 48hr post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | DepoDur80 | DepoDur120 | Control
Number analyzed (Participants) | 6 | 0 | 7
Participants | 1 |  | 1

11. Secondary Outcome: Number of Participants That Were Bradycardia Within 48hr Post Surgery
Description: Number of participants that were bradycardia within 48hr post surgery
Time Frame: 48hr post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | DepoDur80 | DepoDur120 | Control
Number analyzed (Participants) | 6 | 0 | 7
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | DepoDur80 | DepoDur120 | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/0 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/0 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/0 | 0/7

LIMITATIONS AND CAVEATS:
The study was stopped short as the manufacturer decided to stop drug production; therefore without a complete enrollment, statistical analysis was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No